CLINICAL TRIAL: NCT04787926
Title: A Multicenter, Open-Label Study to Evaluate the Safety and Performance of DuraLock-C 4.0%, 30.0%, and 46.7% for the Maintenance of Central Venous Catheter Patency in Adult Hemodialysis Subjects Treated in Clinic
Brief Title: DuraLock-C Catheter Lock Solution
Status: Terminated | Type: Observational
Why Stopped: Enrollment was low or halted with few to zero future anticipated enrollments.
Sponsor: Medical Components, Inc dba MedComp (Industry)
Collaborators: Syneos Health (Other); Veeva Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: 003
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Catheter-Related Infections; Citrate Adverse Reaction
Keywords: Catheter Lock; Trisodium Citrate
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Duralock-C 4%: DuraLock-C 4.0%: Pouch Contains: (2) 3 mL Syringes w/ 2.5 mL Trisodium Citrate Dihydrate 40 mg/mL Solution Contains: Trisodium Citrate Dihydrate, Citric Acid Anhydrous, Water
  Interventions: Device: Locking Solution
- Duralock-C 30%: DuraLock-C 30.0%: Pouch Contains: (2) 3 mL Syringes w/ 2.5 mL Trisodium Citrate Dihydrate 300 mg/mL Solution Contains: Trisodium Citrate Dihydrate, Citric Acid Anhydrous, Water
  Interventions: Device: Locking Solution
- Duralock-C 46.7%: DuraLock-C 46.7%: Pouch Contains: (2) 3 mL Syringes w/ 2.5 mL Trisodium Citrate Dihydrate 467 mg/mL Solution Contains: Trisodium Citrate Dihydrate, Citric Acid Anhydrous, Water
  Interventions: Device: Locking Solution

INTERVENTIONS:
Device: Locking Solution — The total duration of the study treatment period will be 90 calendar days, from Visit 1 Pre-Instillation to the last study-related assessment. Two to 3 instillations (1 per lumen per visit) of DuraLock-C 4.0%, 30.0%, or 46.7% (equivalent to the catheter manufacturer's prescribed priming volume) will be instilled 1 to 3 days apart (with a HD schedule of 3 to 4 times per week); each instillation of CLS will remain in the CVC for approximately 24 to 72 hours ± 12 hours, based on their practice preferences. EOS will take place at the patient's next scheduled dialysis session.

SUMMARY:
To evaluate the safety and performance of DuraLock-C 4.0%, 30.0%, and 46.7% for the maintenance of central venous catheter (CVC) patency in adult hemodialysis (HD) patients

DETAILED DESCRIPTION:
This study is a multicenter, open-label, post-market study to evaluate the safety and performance of DuraLock-C 4.0%, 30.0%, and 46.7% in the maintenance of catheter patency of an indwelling HD CVC in adult HD patients treated in clinic.

On Day 0, patients to be instilled who meet all of the inclusion criteria and none of the exclusion criteria will be enrolled in the study to receive 1 of the 3 DuraLock-C solutions. It is expected that a minimum of 3 sites will enroll patients to the study in order to cover the 3 solutions to be tested; each site will enroll to 1 unique DuraLock-C solution only, until the sample size for the solution has been reached.

DuraLock-C 4.0%, 30.0%, or 46.7% solutions will be instilled to lock the catheter as part of the routine care of the patient. Individual patients will receive the catheter locking solution (CLS) as a catheter lock post-HD session until catheter dysfunction is observed or until the end of the study period (Calendar Day 90). The CLSs are commercially available and will not be provided as part of the study design.

End of Study (EOS) will take place at the patient's next scheduled session.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females will be eligible for study entry provided that all inclusion/exclusion criteria are satisfied.

Patients must fulfill all of the following inclusion criteria to be eligible for participation in the study:

1. Able to give informed consent after an explanation of the proposed study, and who are willing to comply with the study requirements for therapy during the entire study treatment period.
2. Patients undergoing HD 3 or 4 times per week in clinic (expected to continue for the length of the study) with an established or newly placed non-tunneled or tunneled HD CVC as primary vascular access.
3. Adult male or female patients, aged ≥18 years at the time of screening.
4. Clinically stable as judged by the treating physician and as demonstrated by stable medical history for 30 days prior to enrollment, physical examination, and laboratory testing.
5. Expected to survive for the next 6 months and the patient is likely to require the use of a CVC for at least 90 days.
6. Females of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) pregnancy test at screening

Exclusion Criteria:

* 1. Patients with an arteriovenous fistula or arteriovenous graft in use at the time of the study.

  2. Patients with a history of thromboembolic disease. 3. Patients with a history of HD catheter dysfunction due to thrombosis or a blood pump speed rate <300 mL/min during HD in the past 30 days.

  4. Patients with uncontrolled abnormal coagulation parameters and are at additional risk for clotting or excessive bleeding.

  5. Patients who received antibiotics within the last 14 days. 6. Have had an acute infection ≤ 30 days prior to enrollment. 7. Known allergy to heparin, including HIT. 8. Patients who received thrombolytic treatment (ie, tissue plasminogen activator [tPA]) within 4 weeks of enrollment.

  9. Patients using any type of antimicrobial-coated or heparin-coated catheter. 10. Have a positive serology test for human immunodeficiency virus or hepatitis infection.

  11. Current requirement for systemic immunosuppression that would increase risk of infection or any form of immunosuppressive disease.

  12. Patient is currently taking another medication with known systemic drug interaction with citrate or heparin.

  13. Patient is anticipated to receive a renal transplant within the study period should be excluded.

  14. Patients with known or suspected liver failure. 15. Are female and pregnant, lactating, or planning to become pregnant during the study period.

  16. Are currently participating in another interventional clinical study or has participated in another interventional clinical study in the past 3 months or previous enrollment in this study.

  17. Patient has a condition the investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk.

  18. Patient has an active malignancy of any type, or has been diagnosed with cancer within 5 years prior to screening (excluding squamous or basal cell carcinoma of the skin).

  19. Patient has a known allergy or history of significant adverse reaction to trisodium citrate or related compounds or to any of the excipients (citric acid).

  20. Any clinically significant abnormal laboratory test results found during medical screening, as determined by the investigator. NOTE: A test value above or below the normal range does not necessarily indicate that the value is "clinically significant." The determination should be made by the investigator.

  21. Have a history of noncompliance with HD as assessed by an investigator. 22. Have had a major cardiovascular or cerebrovascular event within 3 months of study entry.

  23. Are scheduled for living-donor transplantation within the study period, plan to change to peritoneal dialysis (PD) therapy within the study period, plan to change to a home HD treatment, or plan to relocate to an area where no study center is located.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing hemodialysis (HD) via a central venous cathter (CVC).
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Primary Catheter Patency | 90 days
  Catheter Flow

SECONDARY OUTCOMES:
CRBSI | 90 Days
  Incidence of catheter-related bloodstream infection (CRBSI) over the course of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique HEMERA Pays de Caux, 14 .A avenue Foch, Yvetot, France

IPD SHARING:
Plan to Share IPD: Undecided
Publication undecided